CLINICAL TRIAL: NCT00540176
Title: A Phase II Open-labeled, Double-arm Clinical Study of Dichloroacetate (DCA) in Malignant Gliomas and Glioblastome Multiforme (GBM) Patients
Brief Title: The Safety and Efficacy of DCA for the Treatment of Brain Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Capital Health, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCA 10002
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2010-02

CONDITIONS: Malignant Gliomas, Glioblastoma Multiforme
Keywords: Dichloroacetate; Glioblastoma Multiforme; Glioma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (Experimental): Recurrent disease with previous surgery, radiation therapy and/or chemotherapy
  Interventions: Drug: Dichloroacetate (DCA)
- Cohort B (Experimental): Newly diagnosed disease with no previous therapy
  Interventions: Drug: Dichloroacetate (DCA)

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Oral DCA given twice daily for the 24 week period of the study. Continuation of therapy will be indefinite if efficacious.

SUMMARY:
Malignant gliomas, which include Glioblastoma multiforme (GBM), are the most common and most aggressive types of brain cancer, accounting for approximately 60% of primary brain tumors. These tumors are characterized by diverse molecular abnormalities (within the same tumor), which, along with the difficulties of many standard chemotherapies crossing the blood barrier, contribute to the very poor response to therapy and poor survival.

We recently showed that Dichloroacetate (DCA, an inhibitor of the mitochondrial pyruvate dehydrogenase kinase) was able to depolarize cancer (but not normal) mitochondria and induce apoptosis in cancer but not normal tissues. We believe that altering the metabolism of cancers like glioblastoma (DCA switches metabolism from the cytoplasmic glycolysis to the mitochondrial glucose oxidation) we inhibit the resistance to apoptosis that characterizes cancer. Because metabolism (i.e. glycolysis) is the end result of many and diverse molecular pathways, the effects of DCA might be positive in cancers with diverse molecular backgrounds. DCA is also a very small molecule that readily crosses the blood brain barrier. Therefore we hypothesize that DCA will be an effective and relative non-toxic potential therapy for malignant gliomas.

We are conducting a phase II trial with 2 parallel arms: a) patients with newly diagnosed malignant gliomas and b) patients with recurrent gliomas or gliomas that have failed standard therapy (which includes surgery, radiotherapy and chemotherapy). All patients need to have a histological diagnosis. DCA will be given orally and patients will be followed for a minimum of 6 months. The tumor size will be followed by standard MRI or CT criteria and glucose uptake (a direct effect of DCA on the tumor) will be measured by FDG-PET imaging. Several clinical parameters and quality of life will be followed. Potential toxicity (particularly peripheral neuropathy) will be closely followed and dose-de-escalation protocols are in place in case of toxicity. In addition, escape protocols for the application of standard therapy (when appropriate) are in place in patients with no evidence of response to DCA. In vitro studies will be performed in the tissues obtained at the time of surgery (where appropriate) and correlated prospectively with clinical data.

There is limited ability to accept patients outside of Alberta; this is in part because the visit and testing schedule is intense, requiring residence in Edmonton for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed intracranial malignant glioma / GBM tumors.
* All patients enrolled must have measurable with or without evaluable disease, as defined in Section 11.
* In the recurrent malignant glioma cohort of patients, four weeks must have elapsed from prior chemotherapy or radiation therapy.
* Age 18 years and over.
* ECOG (Eastern Cooperative Oncology Group) performance status Grade 0-2 (Karnofsky >70).
* Life expectancy of greater than 12 weeks.
* Patients must have liver, kidney and marrow function as defined below:

  * absolute neutrophil count >1,500/mcL
  * hemoglobin >90 g/L
  * platelets >100,000/mcL
  * total bilirubin <1.5 X upper limit of normal (ULN)
  * AST(SGOT) and ALT(SGPT) <1.5 X ULN
  * creatinine <1.5 X ULN
* Recovery to baseline or, at most, grade 1 of all drug-related toxicities due to prior chemotherapy, radiation, or molecular targeted therapy, except for alopecia.
* Women of child-bearing potential and men must agree to use adequate contraception (e.g.: hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria

* Patients who have had chemotherapy, molecular targeted therapy, or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with new onset or increasing dose regimen of steroids for the week prior to enrollment.
* Patients cannot be receiving any other investigational therapies.
* Patients with grade 2 or higher peripheral neuropathy due to prior medical condition (such as multiple sclerosis, diabetes etc), medications (chemotherapy), or other etiologies.
* Greater than 0.8 cm brain midline shift on CT scan or MRI
* Any psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes with history of significant hypoglycemic episodes in the past 3 months or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with DCA. In addition, these patients are at increased risk of lethal (and at time intracranial) infections when treated with potentially marrow-suppressive therapy.
* History of malabsorption syndrome or substantial amount of small bowels or stomach resection or obstruction that may impair absorption of DCA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine the therapeutic response to oral Dichloroacetate (DCA) in patients with malignant gliomas, utilizing standard criteria for the objective response of tumor size to treatment (CT and/or MRI).
To evaluate the safety and tolerability of oral (DCA) in patients with gliomas.
To determine the progression-free survival (PFS) and overall survival achieved with oral DCA in patients with gliomas.

SECONDARY OUTCOMES:
• To evaluate the in vitro effects of DCA on cell proliferation/apoptosis and mitochondrial function in malignant glioma tissues taken from enrolled patients at the time of surgery and correlate them with clinical data.
• To evaluate glucose uptake using 18F-FDG Positron Emission Tomography (PET) scanning as a biological marker for predicting subsequent therapeutic response to oral DCA in patients with malignant gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Petruk, MD co-PI, Principal Investigator — University of Alberta and Capital Health; Evangelos D Michelakis, MD co-PI, Principal Investigator — University of Alberta and Capital Health; Connor Maguire MD, investigator, Principal Investigator — University of Alberta and Capital Health; Linda Webster, NP manager, Study Director — Capital Health, Canada
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Bonnet S, Archer SL, Allalunis-Turner J, Haromy A, Beaulieu C, Thompson R, Lee CT, Lopaschuk GD, Puttagunta L, Bonnet S, Harry G, Hashimoto K, Porter CJ, Andrade MA, Thebaud B, Michelakis ED. A mitochondria-K+ channel axis is suppressed in cancer and its normalization promotes apoptosis and inhibits cancer growth. Cancer Cell. 2007 Jan;11(1):37-51. doi: 10.1016/j.ccr.2006.10.020. PMID 17222789